CLINICAL TRIAL: NCT06451809
Title: Prediction of the Response to a Course of Transcranial Magnetic Stimulation (rTMS) Based on the Acute Variation in Heart Rate Variability Obtained After a Single RTMS Session in Patients with Major Depressive Disorder
Brief Title: Prediction of the Response to a Course of Transcranial Magnetic Stimulation (rTMS) Based on Heart Rate Variability
Acronym: DEP&MOD
Status: Suspended | Type: Observational
Why Stopped: We are faced with a decrease in rTMS activity at the study sites, as well as problems with the active file meeting the protocol inclusion criteria, resulting in a low recruitment rate and an extended study timetable, forcing us to suspend this study.
Sponsor: GCS CIPS (Other)
Responsible Party: Sponsor
Other Study IDs: DEP&MOD
Record Dates: First submitted 2024-05-29; First posted 2024-06-11 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with MDD: Patients who are prescribed a course of 30 rTMS sessions to treat an episode of MDD at one of the nine participating centres
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — rTMS will be applied 5 days out of 7 for 6 weeks, for a total of 30 sessions. The area stimulated will be the left dorsolateral prefrontal cortex, at a frequency of 10 Hz, at 110% of motor threshold for approximately 20 minutes (i.e. 3,000 stimulations per session).

SUMMARY:
Changes in heart rate variability following a single session of rTMS will be tested as a predictor of response to a course of 30 rTMS sessions in patients with major depressive disorder (MDD).

DETAILED DESCRIPTION:
The objective of this study is to investigate whether acute changes in heart rate variability following a single session of repetitive transcranial magnetic stimulation (rTMS) can predict the response to a 30-session course of rTMS in patients with major depressive disorder (MDD) with good sensitivity and specificity. Patients who are prescribed rTMS to treat an episode of MDD at one of the nine participating centres will be invited to participate in the study. The protocol includes one inclusion visit and seven evaluation visits before, during, and after the course of rTMS. The rTMS course will last for six weeks, comprising of 30 sessions with five sessions per week. Prior to the start of the rTMS course, the patient will have to fill in a number of questionnaires. Before the first session, heart rate variability will be assessed by recording the RR interval at rest using a heart rate belt on the armchair stimulation. A second RR interval recording will be taken immediately after the first rTMS session. Patients will answer questionnaires weekly and after the final rTMS session to track the progression of depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Having a prescription for a course of rTMS to treat an episod of MDD
* Unipolar MDD confirmed according to DSM-5 criteria
* Moderate to severe MDD (MADRS score > 19)
* No use of psychotropic medication or use stabilised (no change in dose < 4 weeks before study entry)
* Able to understand, speak, read and write French
* Express informed consent, after a period of reflection
* Affiliated with a French social security scheme or beneficiary of such a scheme

Exclusion criteria:

* History of epilepsy or convulsive seizures
* Previous brain surgery
* History of recent cranial trauma (< 6 months)
* Presence of severe suicidal ideation
* Psychotic disorders
* Metal objects in the head, eyes or brain
* Implanted ferromagnetic equipment (pace maker, cochlear implant, etc.)
* Clinical evidence of serious or uncontrolled alcohol or substance use disorders in the three months prior to the study
* Active withdrawal from alcohol or other substances
* One or more recent rTMS sessions (< 4 weeks)
* Other non-drug therapy recently initiated (< 4 weeks) to treat MDD (psychotherapy, phototherapy, vagus nerve stimulation, etc.)
* Prescription of cardiotropic drugs belonging to the following classes: predominantly cardiac calcium channel blockers, Vaughan Williams class I anti-arrhythmics and beta-blockers.
* Subjects in a period of relative exclusion from another protocol
* Adults protected by law or patients under guardianship or curatorship
* Subjects deprived of their liberty by judicial or administrative decision
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited will be patients who have been admitted as an outpatient for the treatment of MDD by rTMS treatment at one of the 9 study centres.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Threshold of variation in terms of RMSSD between normal heartbeats enabling to predict the response to the course of rTMS with the best possible sensitivity and specificity. | One day for heart rate variability records (Before and after the first rTMS session), and 6 weeks for assessing the MADRS scores (before and after the course of 30 rTMS sessions)
  Threshold of variation in terms of RMSSD (root mean square of successive differences) between normal heartbeats after a single rTMS session enabling to predict the response to the course of rTMS with the best possible sensitivity and specificity. The response to the course of rTMS will be assessed via the evolution of the MADRS score (decrease of MADRS score >50%)

SECONDARY OUTCOMES:
Threshold of other heart rate variability markers enabling to predict the response to the course of rTMS with the best possible sensitivity and specificity. | One day for heart rate variability records (Before and after the first rTMS session), and 6 weeks for assessing the MADRS scores (before and after the course of 30 rTMS sessions)
  Threshold of variation in other heart rate variability markers (SDNN, low frequencies, high frequencies and low to high frequencies ratio) after a single rTMS session enabling to predict the response to the course of rTMS with the best possible sensitivity and specificity. The response to the course of rTMS will be assessed via the evolution of the MADRS score (decrease of MADRS score >50%)
Threshold of variation in heart rate variability markers enabling to predict the remission to the course of rTMS with the best possible sensitivity and specificity. | One day for heart rate variability records (Before and after the first rTMS session), and 6 weeks for assessing the MADRS scores (before and after the course of 30 rTMS sessions)
  Threshold of variation in heart rate variability markers (RMSSD, SDNN, low frequencies, high frequencies and low to high frequencies ratio) after a single rTMS session enabling to predict the remission to the course of rTMS with the best possible sensitivity and specificity. The remission to the course of rTMS will be assessed via the evolution of the MADRS score (MADRS ≤ 10 after the course of rTMS)

OTHER OUTCOMES:
Self-evaluation of depressive symptoms | 6 weeks (baseline and weekly records)
  PHQ9 questionnaire
Sleep quality | 6 weeks (baseline and after the course of 30 rTMS sessions)
  PSQI questionnaire
Physical activity and sedentary behaviors | 6 weeks (baseline and after the course of 30 rTMS sessions)
  SIMPAQ questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Kabirian, MD, Principal Investigator — France Chief Medical Officer, Clariane
Locations (9):
- France (9):
  - Clinique Inicea du Pays de Seine, Bois-le-Roi
  - Clinique Inicea La Mare O Dans, Les Damps
  - Clinique Inicea Villa des Roses, Lyon
  - Etablissement public de santé de Ville-Evrard, Neuilly-sur-Marne
  - Centre médical de psychiatrie NeuroStim Luxembourg, Paris
  - Centre médical de psychiatrie NeuroStim Etoile, Paris
  - Clinique Inicea Jeanne d'Arc Hopital Privé Parisien, Saint-Mandé
  - Centre montois de psychiatrie ambulatoire Inicea, Saint-Pierre-du-Mont
  - Centre Tourangeau de psychiatrie ambulatoire Inicea, Tours

IPD SHARING:
Plan to Share IPD: Undecided